CLINICAL TRIAL: NCT00680095
Title: 21-day Cumulative Irritation Test
Brief Title: Cumulative Irritation Test
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Other
Other Study IDs: AN2690-ONYC-101; C3371011 (Other: Alias Study Number)
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Onychomycosis
Keywords: Onychomycosis; Fungal Nail
MeSH Terms: conditions — Onychomycosis | interventions — tavaborole; Sodium Dodecyl Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- A (Experimental): AN2690 Solution, 2.5%
  Interventions: Drug: AN2690
- B (Experimental): AN2690 Solution, 7.5%
  Interventions: Drug: AN2690
- C (Experimental): AN2690 Solution, 5.0%
  Interventions: Drug: AN2690
- D (Active Comparator): AN2690 Solution, Vehicle
  Interventions: Other: AN2690 Solution, Vehicle
- E (Active Comparator): Sodium Lauryl Sulfate, 0.5%
  Interventions: Other: Sodium Lauryl Sulfate, 0.5%

INTERVENTIONS:
Drug: AN2690 — AN2690 Solution, 2.5%, Daily for up to 21 days
  Arms: A
Drug: AN2690 — AN2690 Solution, 7.5%, Daily for up to 21 days
  Arms: B
Drug: AN2690 — AN2690 Solution, 5.0%, Daily for up to 21 days
  Arms: C
Other: AN2690 Solution, Vehicle — AN2690 Solution, Vehicle, Daily for up to 21 days
  Arms: D
Other: Sodium Lauryl Sulfate, 0.5% — Sodium Lauryl Sulfate, 0.5%, Daily for up to 21 days
  Arms: E

SUMMARY:
The purpose of this study is to determine the cumulative irritation potential of the products listed by the Sponsor.

DETAILED DESCRIPTION:
Healthy, adult volunteers of either sex will be patched on his/her back with AN2690 Solution 2.5%, AN2690 Solution 5%, AN2690 Solution 7.5%, AN2690 Solution Vehicle and Sodium Laurel Sulfate 0.5% over the course of 21 consecutive days. After 24 hours, the patches are to be removed and the site evaluated using a five-point scale for irritation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, volunteers of either sex, at least 18 years of age or older
* Females of childbearing potential submitted to a urine pregnancy test and had negative results at Day 1 and at the final visit and also was using an effective method of birth control (e.g. abstinence, implants, injectables, oral contraceptives, intrauterine contraceptive devices or double barrier) or agreed to use an effective method of birth control prior to becoming sexual active
* Subjects were of any skin type or race providing their degree of pigmentation did not interfere with making readings of skin reactions
* Subjects were willing to follow the study procedures and complete the study
* Written informed consent was obtained

Exclusion Criteria:

* Subject with any skin disease that would have in any way confounded interpretation of the study results. Atopic dermatitis/eczema, psoriasis or chronic asthma were excluded
* Subject was pregnant or nursing
* Subject had a history of sensitivity to any component of any of the formulations
* Use of chronic medications (such as antihistamines, corticosteroids, analgesics and anti-inflammatories) for one week before and during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-01-22 (Actual); Primary Completion 2007-02-19 (Actual); Study Completion 2007-02-19 (Actual)

PRIMARY OUTCOMES:
Severe irritation (Grade 3 or 4) observed at any site | Daily for 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- The Education and Research Foundation, Inc., Lynchburg, Virginia, United States